CLINICAL TRIAL: NCT00605969
Title: Hip Reconstruction and Modeling for Surgical Pre-Operative Planning
Brief Title: Dynamic Imaging of the Hip for Pre-operative Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2006-552
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Femoroacetabular, Impingement
Keywords: femoroacetabular, impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAI patients (Active Comparator): This group consists of participants diagnosed with femoroacetabular impingement that are undergoing surgical correction.
  Interventions: Procedure: Motion analysis; Diagnostic Test: Computed Tomography
- Control (Placebo Comparator): This group consists of healthy control participants with no hip problems.
  Interventions: Procedure: Motion analysis; Diagnostic Test: Computed Tomography

INTERVENTIONS:
Procedure: Motion analysis — Participants will undergo a motion analysis procedure: a dynamic assessment of the movement in their hip.
Diagnostic Test: Computed Tomography — Participants will undergo computed tomography (CT) scan of their hip.

SUMMARY:
One of the leading causes of hip arthritis is femoro-acetabular impingement which means the hip joint is deformed such that the hip joint jams in the front when the hip is bent all the way forward. This can lead to significant damage to the hip joint and may result in the need for a total hip replacement. However, if detected early, this deformity can be treated surgically by reshaping the hip joint. If the hip joint could be better visualized before surgery, then surgeons would be able to develop less invasive surgical techniques to correct this deformity.

DETAILED DESCRIPTION:
In this study, we are trying to develop a way to help surgeons visualize the hip joint before surgery in order to assist with pre-operative planning. This will be done by comparing the dynamic hip images in patients with femoroacetabular impingement to the hip images of healthy volunteers with no hip problems.

ELIGIBILITY:
Inclusion Criteria:

* All participants (patients and controls) must be between the ages of 18 and 55, with a BMI less than 35.

The patients must have a probable diagnosis of femoro-acetabular impingement (FAI). Their hip pain must have been ongoing for at least 3 months. The controls must have a normal hip as defined by AP pelvis radiographs.

Exclusion Criteria:

* Participants (patients and controls) will be excluded if they are pregnant, have a knee injury or replacement, or history of childhood hip disease. Patients will be excluded if have they have arthritis, previous fracture or trauma to the hip, previous hip surgery, dysplasia, or avascular necrosis. Controls will be excluded if they have hip pain.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Validation of kinematic model of hip joint | Within 6 months of recruitment
  Development of a kinematical model of the hip joint to simulate virtual joint motion. This will be done by using automatic segmentation using the CT data to generate models.

SECONDARY OUTCOMES:
Joint Kinetics | 24 months
  Retro-reflective markers will be placed on each participant in a laboratory setting. Joint kinematics will be reconstructed from marker trajectories recorded by a camera system. Together, with EMG data, the investigators will calculate joint kinetics
Muscle Activity | 24 months
  Retro-reflective markers will be placed on each participant in a laboratory setting. Electromyography (EMG) electrodes will be placed on the skin above the tibialis anterior, medial and lateral gastrocnemius, vastus lateralis and medialis, biceps femoris, semitendinosis and gluteus maximums of both limbs. Muscle activity will be measured using EMG signal recorded during activity.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaule, MD, FRCSC, Principal Investigator — University of Ottawa / The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Ng KC, Lamontagne M, Adamczyk AP, Rakhra KS, Beaule PE. Patient-specific anatomical and functional parameters provide new insights into the pathomechanism of cam FAI. Clin Orthop Relat Res. 2015 Apr;473(4):1289-96. doi: 10.1007/s11999-014-3797-1. PMID 25048279
- [Result] Kennedy MJ, Lamontagne M, Beaule PE. Femoroacetabular impingement alters hip and pelvic biomechanics during gait Walking biomechanics of FAI. Gait Posture. 2009 Jul;30(1):41-4. doi: 10.1016/j.gaitpost.2009.02.008. PMID 19307121
- [Result] Lamontagne M, Kennedy MJ, Beaule PE. The effect of cam FAI on hip and pelvic motion during maximum squat. Clin Orthop Relat Res. 2009 Mar;467(3):645-50. doi: 10.1007/s11999-008-0620-x. Epub 2008 Nov 26. PMID 19034598
- [Result] Lamontagne M, Brisson N, Kennedy MJ, Beaule PE. Preoperative and postoperative lower-extremity joint and pelvic kinematics during maximal squatting of patients with cam femoro-acetabular impingement. J Bone Joint Surg Am. 2011 May;93 Suppl 2:40-5. doi: 10.2106/JBJS.J.01809. PMID 21543687
- [Result] Brisson N, Lamontagne M, Kennedy MJ, Beaule PE. The effects of cam femoroacetabular impingement corrective surgery on lower-extremity gait biomechanics. Gait Posture. 2013 Feb;37(2):258-63. doi: 10.1016/j.gaitpost.2012.07.016. Epub 2012 Aug 28. PMID 22939410